CLINICAL TRIAL: NCT00122317
Title: Open Label Extension Study of Eculizumab in Patients With Transfusion Dependent PNH
Brief Title: Extension Study of Eculizumab in Patients With Transfusion Dependent Paroxysmal Nocturnal Hemoglobinuria (PNH)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E05-001
Record Dates: First submitted 2005-07-20; First posted 2005-07-22 (Estimated); Results first posted 2017-06-05 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2018-02

CONDITIONS: Paroxysmal Hemoglobinuria, Nocturnal
Keywords: transfusion dependent; paroxysmal nocturnal hemoglobinuria; hemolytic
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal; Hemolysis | interventions — eculizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Eculizumab (Experimental): 600 mg intravenous infusion every week x 4 then 900 mg iv every two weeks
  Interventions: Drug: eculizumab

INTERVENTIONS:
Drug: eculizumab
  Other Names: Soliris

SUMMARY:
The purpose of this study is to evaluate the long-term safety of eculizumab in patients with transfusion dependent hemolytic PNH.

DETAILED DESCRIPTION:
An open-label extension study to evaluate long-term safety of eculizumab in PNH patients who had completed the TRIUMPH (C04-001), SHEPHERD (C04-002), and X03-001 studies.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have fully completed the TRIUMPH, SHEPHERD, or X03-001 studies
* TRIUMPH patients who have discontinued receiving investigational drug prior to the last visit of the study due to lack of efficacy or exacerbation of symptoms of PNH and have completed all monthly safety and efficacy procedures
* Patient must be willing and able to give written informed consent
* Patient must avoid conception during the trial

Exclusion Criteria:

* Patients who have terminated early from the SHEPHERD or X03-001 studies
* Patients who have terminated early from the TRIUMPH study due to an adverse event
* Female who is pregnant, breast feeding, or intending to conceive during the course of the study
* Any condition that could increase the patient's risk by participating in the study or could confound the outcome of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2005-05 (Actual); Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (40):
- United States (14):
  - Stanford University Medical Center, Division of Hematology, Stanford, California
  - Hartford Hospital, Cancer Clinical Research Office, Hartford, Connecticut
  - Cleveland Clinic Florida, Department of Clinical Research, Weston, Florida
  - Indianapolis University Cancer Center, Indianapolis, Indiana
  - Johns Hopkins University Medical Center, Baltimore, Maryland
  - National Heart, Lung, and Blood Institute, National Institutes of Health, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic, Divison of Hematology, Rochester, Minnesota
  - Washington University, Department of Internal Medicine/Division of Hematology, St Louis, Missouri
  - NYU Clinical Cancer Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Division Cell Therapy, Heme Malignancies Program, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Presbyterian Medical Center, PENN Comprehensive Hemophilia & Thombosis Program, Philadelphia, Pennsylvania
- Australia (5):
  - Royal North Shore Hospital, Haematology Department, Saint Leonards, New South Wales
  - Princess Alexandra Hospital, Oncology Haematology Radiation Department, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Haematology/Oncology Department, Woodville South, South Australia
  - The Royal Perth Hospital, Department of Haematology/Level 2, Perth, Western Australia
  - Royal Melbourne Hospital, Department of Clinical Haematology & Medical Oncology, Parkville
- Ucl St. Luc, Hematology Department, Brussels, Belgium
- Canada (2):
  - University of Alberta, Cross Cancer Institute, Edmonton, Alberta
  - London Regional Cancer Centre, Clinical Research Unit Room C3080, London, Ontario
- Hopital Saint Louis, Centre d'investigation Clinique, Paris, Cedex, France
- Germany (4):
  - Universitatsklinikum Essen, Zentrum fur Innere Medizin, Essen
  - Medizinische Hochschule Hannover, Abt. Hamatologie/Onkologie, Zentrum fur Innere Medizin, Hanover
  - Universitatskliniken des Saarlandes, Innere Medizin 1, Homburg/Saar
  - Institut fur Klinische Transfusionmedizin und Immunogenetik, Abtlg. Transfusionmedizin des Univ. Ulm, Ulm
- St. James's Hospital, Cancer Clinical Trial Office, Dublin, Ireland
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Dipartimento di area critica medico-chirurgica, Florence
  - Ospedale San Martino, Department of Hematology, Genova
  - Ospedale Maggiore di Milano, Divisione di Ematologia, Milan
  - Universita degli Studi di Napoli, Divisione di Ematologia, Azienda Universitar Policlinico, Napoli
  - Ospedale San Bortolo, Divisione di Ematologia, Vicenza
- UMC St. Radboud, Department of Hematology, Nijmegen, GA, Netherlands
- Spain (3):
  - Hospital Clinic i Provincial, Servicio de Hematologia, Barcelona
  - Hospital Universitario Germans Trias I Pujol, Servicio de Hematologia, Barcelona
  - Hospital De La Paz, Servicio de Hematologia, Madrid
- Stockholm South Hospital, Division of Hematology, Stockholm, Sweden
- United Kingdom (2):
  - Leeds General Infirmary, D Floor Brotherton Wing, Leeds
  - St. George's Hospital, Department of Haematology, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillmen P, Muus P, Duhrsen U, Risitano AM, Schubert J, Luzzatto L, Schrezenmeier H, Szer J, Brodsky RA, Hill A, Socie G, Bessler M, Rollins SA, Bell L, Rother RP, Young NS. Effect of the complement inhibitor eculizumab on thromboembolism in patients with paroxysmal nocturnal hemoglobinuria. Blood. 2007 Dec 1;110(12):4123-8. doi: 10.1182/blood-2007-06-095646. Epub 2007 Aug 16. PMID 17702897

RESULTS

PARTICIPANT FLOW:
Groups:
- Eculizumab: eculizumab: 600 mg intravenous infusion every week x 4 then 900 mg iv every two weeks
Period: Overall Study
Arm/Group | Eculizumab
Started | 187
Completed | 176
Not Completed | 11
Not completed — Death | 3
Not completed — Adverse Event | 4
Not completed — Physician Decision | 2
Not completed — patient non-compliance | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Eculizumab
Number analyzed (Participants) | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.1 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101
  Male | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 6
  Black | 7
  Caucasian | 168
  Other | 6

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment-emergent Adverse Events
Time Frame: From time of consent to a maximum of 2.5 years of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Eculizumab
Number analyzed (Participants) | 187
Participants | 182

2. Secondary Outcome: Hemolysis as Measured by Change From Baseline in LDH Area Under the Curve
Time Frame: From time of first infusion through 24 months of study treatment
Measure: Mean (Standard Deviation); unit: U/L x Day
Arm/Group | Eculizumab
Number analyzed (Participants) | 184
U/L x Day | -365185.8 (210407.1)

3. Secondary Outcome: Quality of Life as Measured by FACIT-Fatigue Scale Change From Baseline
Description: The FACIT-Fatigue scale is a collection of quality of life questionnaires pertaining to the management of fatigue symptoms due to a chronic illness. The FACIT-Fatigue is a 13-item questionnaire that assesses self-reported fatigue and its impact upon daily activities and function over the preceding 7 days. Patients score each item on a 5-point scale: 0 (Not at all) to 4 (Very much). Total scores range from 0 to 52, with higher score indicating better quality of life.
Time Frame: From time of first infusion through 24 months of study treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eculizumab
Number analyzed (Participants) | 184
units on a scale | 9.24 (12.42)

4. Secondary Outcome: Incidence of Thrombosis After Eculizumab Infusion
Description: Thrombosis was defined as occurrence of major adverse vascular events
Time Frame: From time of first ever dose through last dose (up to 24 months of study treatment)
Measure: Number; unit: Number of events per 100 patient-years
Arm/Group | Eculizumab
Number analyzed (Participants) | 184
Number of events per 100 patient-years
  Prior to first eculizumab dose | 7.82
  From first dose of eculizumab through last dose | 1.99

ADVERSE EVENTS:
Time Frame: From time of consent to a maximum of 2.5 years of study treatment
Arm/Group | Eculizumab
All-Cause Mortality (participants affected / at risk) | 3/187
Serious Adverse Events (participants affected / at risk) | 57/187
Other Adverse Events (participants affected / at risk) | 180/187
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=187)
Agranulocytosis (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Aplastic anaemia (Blood and lymphatic system disorders) | 2
Haemolysis (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 1
Paroxysmal Nocturnal Haemoglobinuria (Renal and urinary disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Cardiac Failure (Cardiac disorders) | 1
Retinal vein thrombosis (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 5
Ascites (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Sigmoiditis (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Pyrexia (General disorders) | 5
Bile duct stone (Hepatobiliary disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 3
Cholecystitis acute (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Hepatic vein thrombosis (Hepatobiliary disorders) | 1
Portal vein thrombosis (Hepatobiliary disorders) | 2
Bacterial sepsis (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Cellulitis gangrenous (Infections and infestations) | 1
Empyema (Infections and infestations) | 1
Endocarditis (Immune system disorders) | 1
Enterococcal sepsis (Infections and infestations) | 1
Gallbladder abscess (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 2
Haemophilus infection (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 2
Meningococcal sepsis (Infections and infestations) | 2
Necrotising fasciitis (Infections and infestations) | 1
Penile infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Respiratory tract infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Staphylococcal Infection (Infections and infestations) | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Viral Infection (Infections and infestations) | 3
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1
Drug Toxicity (Injury, poisoning and procedural complications) | 1
Wrist Fracture (Injury, poisoning and procedural complications) | 1
Haemoglobin Decreased (Investigations) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis Stenosans (Musculoskeletal and connective tissue disorders) | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Chronic Myelomonocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to Bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral Haemorrhage (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Metabolic Encephalopathy (Nervous system disorders) | 1
Suicidal Ideation (Psychiatric disorders) | 1
Calculus Urinary (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 2
Renal Failure Acute (Renal and urinary disorders) | 2
Renal Impairment (Renal and urinary disorders) | 1
Erectile Dysfunction (Reproductive system and breast disorders) | 1
Ovarian Cyst Ruptured (Reproductive system and breast disorders) | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
Phlebothrombosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eculizumab (N=187)
Diarrhoea (Gastrointestinal disorders) | 44
Nausea (Gastrointestinal disorders) | 39
Vomiting (Gastrointestinal disorders) | 38
Abdominal Pain (Gastrointestinal disorders) | 25
Abdominal Pain Upper (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 16
Dyspepsia (Gastrointestinal disorders) | 14
Influenza like Illness (General disorders) | 29
Pyrexia (General disorders) | 18
Oedema Peripheral (General disorders) | 12
Fatigue (General disorders) | 11
Chest Pain (General disorders) | 10
Nasopharyngitis (Infections and infestations) | 74
Upper Respiratory Tract Infection (Infections and infestations) | 58
Urinary Tract Infection (Infections and infestations) | 20
Viral Infection (Infections and infestations) | 17
Sinusitis (Infections and infestations) | 15
Gastroenteritis (Infections and infestations) | 12
Herpes Simplex (Infections and infestations) | 12
Bronchitis (Infections and infestations) | 10
Influenza (Infections and infestations) | 10
Contusion (Injury, poisoning and procedural complications) | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 33
Back Pain (Musculoskeletal and connective tissue disorders) | 32
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 25
Myalgia (Musculoskeletal and connective tissue disorders) | 17
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 61
Dizziness (Nervous system disorders) | 21
Insomnia (Psychiatric disorders) | 11
Cough (Respiratory, thoracic and mediastinal disorders) | 29
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 25
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14
Rash (Skin and subcutaneous tissue disorders) | 12
Pruritus (Skin and subcutaneous tissue disorders) | 11
Haematoma (Vascular disorders) | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Participation in this multicenter study involved a commitment to publish the data from the study in a cooperative publication prior to release of study results on an individual basis.